CLINICAL TRIAL: NCT04599673
Title: Prospective Analysis of Intraoperative AMNIOGEN® Injection in Patients With Rotator Cuff Tear
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yi Ping Wei, Orthopaedic, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-CT7-30(200527-1)
Record Dates: First submitted 2020-09-13; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMNIOGEN (Experimental): Intraoperative1 kit of AMNIOGEN injection into shoulder joint after RCT repair.
  Interventions: Drug: AMNIOGEN
- Normal saline (Placebo Comparator): Intraoperative 10 ml of normal saline injection into shoulder joint after RCT repair.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: AMNIOGEN — AmnioGen® amnion matrix allograft is a bioactive tissue matrix processed from 100% human amniotic tissue. The allograft is processed with advanced technology so the graft can be suspended in liquids and applied through needles and syringes.
  Amniotic tissue is composed of structural extracellular matrix, which is rich in various types of collagen, growth factors, cytokines, and specialized proteins. Thus, the application of amniotic tissue is known to modulate localized tissue inflammation, reduce scar tissue formation and promote the healing of soft tissue.
  Arms: AMNIOGEN
Other: normal saline — 10 ml normal saline
  Arms: Normal saline

SUMMARY:
Purpose: The purpose of this article is to examine the clinical application of AMNIOGEN® in patients with rotator cuff tear.

Methods:

The study was conducted on 100 adult participants with age over affected by unilateral shoulder rotator cuff tear and receiving RCT repair. The investigators divided the participants in two groups, and the group A was treated with perioperative injection of AMNIOGEN® A, group B with perioperative normal saline.

Follow-up:

Every 1,3,and 12months, the investigators recheck physical exmianation at OPD and recheck MRI at postoperative 3 months.

ELIGIBILITY:
Inclusion Criteria:

* receiving unilateral shoulder RCT repair in our hospital postoperative follow-up over 3 month

Exclusion Criteria:

* postoperative follow-up less than 3 month possible pregnency with coagulation disease NSAIDs intake during study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
100 of participants with preoperative and postoperative physical examination are accessed by Empty can test | postoperative 1 month
  the investigators recheck physical exmianation of participants at OPD; physical examination was checked by one orthopedist
100 of participants with preoperative and postoperative physical examination are accessed by Empty can test | postoperative 3 month
  the investigators recheck physical exmianation of participants at OPD; physical examination was checked by one orthopedist
100 of participants with preoperative and postoperative physical examination are accessed by Empty can test | postoperative 12 month
  the investigators recheck physical exmianation of participants at OPD; physical examination was checked by one orthopedist
100 of participants with preoperative and postoperative Magnetic Resonance Imaging are accessed | postoperative 3 month
  size and site of rotator cuff tear was accessed by MRI T1 and T2 image; MRI was checked by one orthopedist

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ping Wei, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Yi Ping Wei, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No